CLINICAL TRIAL: NCT04748549
Title: Intraoperative Virtual Reality for Older Patients Undergoing Total Knee Arthroplasty
Brief Title: Intraoperative VR for Older Patients Undergoing TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Israel-United States Binational Industrial Research and Development Foundation (Unknown); XRHealth (Unknown)
Responsible Party: Principal Investigator, Brian O'Gara, Assistant Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P001176
Record Dates: First submitted 2021-01-29; First posted 2021-02-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Total Knee Arthroplasty
Keywords: Virtual Reality

STUDY DESIGN:
Intervention Model Description: Research participants will be randomized to one of three groups (2:2:1 allocation):
  1. Immersive VR group
  2. Music group
  3. Sham VR + usual care control
  The first 6 patients enrolled will be assigned to the VR group for the purposes of a pilot phase with the objective of identifying and refining any issues with the intervention. Data for these patients will not be included in the statistical analysis.
Who Masked: Outcomes Assessor
Masking Description: Assessors of the Confusion Assessment Method (CAM) and Montreal Cognitive Assessment (MoCA) will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Immersive VR group (Experimental): Patients in the Immersive VR group will don a VR headset connected to a software platform on a tablet, as well as noise cancelling headphones. Patients can choose their desired experience within the VR software from a selection of immersive environments and/or video content. Examples include sitting in a canoe on a river, on a peaceful meadow or in a forest. Patients also have the option to listen to guided meditation or select from a library of videos to watch on a web-based user interface.
  To reduce the influence of the anesthesia provider on the determination of sedative requirements, patients will administer their own sedation according to their needs for relaxation and comfort using a patient controlled system.
  Interventions: Other: Virtual Reality Immersive Relaxation
- Music group (Active Comparator): Patients randomized to the Music group will be equipped with VR headsets but won't view any content. They will also be equipped with noise cancelling headphones in the same fashion as the immersive VR group. A study team member will play from a library of music or other audible content (audiobook, podcast) that was preselected by the patient. Patients in the Sham VR group will also use patient controlled sedation.
  Interventions: Other: Immersive Audio Experience
- Sham VR + Usual Care Control Group (Sham Comparator): Subjects in the control group will wear VR headsets and headphones but will not view any content or listen to any audible content. They will undergo Monitored Anesthesia Care (MAC) according to a prespecified protocol targeting light or moderate sedation with a propofol infusion.
  Interventions: Other: Sham Virtual Reality Experience

INTERVENTIONS:
Other: Virtual Reality Immersive Relaxation — The VR software developed allows patients to select from scenery such as mountains, the beach or from a selection of short videos, which are intended to promote relaxation.
  Arms: Immersive VR group
Other: Immersive Audio Experience — A study team member will play from a library of music or other audible content (audiobook, podcast) that was preselected by the patient.
  Arms: Music group
Other: Sham Virtual Reality Experience — Subjects will wear VR headsets and headphones but will not view any content or listen to any audible content.
  Arms: Sham VR + Usual Care Control Group

SUMMARY:
The objective of this study is to investigate whether the use of virtual reality (VR) during total knee arthroplasty (TKA) can facilitate reductions in intraoperative sedative requirements while maintaining high levels of patient satisfaction as compared to both a music and sham VR + usual care control.

DETAILED DESCRIPTION:
The investigators will conduct a three-armed randomized controlled trial with the following aims:

Specific Aim 1: Evaluate whether the use of VR during TKA can facilitate a reduction in intraoperative propofol dose required for patient comfort as compared to music and sham VR + usual care controls.

Hypotheses: Patients in both the VR and music groups will demonstrate reductions in propofol dose compared to sham VR + usual care controls. A reduction in propofol dose between the VR and music group will be smaller in magnitude.

Specific Aim 2: Assess the effect of VR during TKA on patient reported outcomes including overall satisfaction, pain, and anxiety as compared to music and sham VR + usual care controls.

Hypotheses: Patients in the VR group will report significantly higher satisfaction and better control of pain and anxiety than those in the music group and usual care group.

Specific Aim 3: Explore the potential effects of VR during TKA on other key secondary outcomes of perioperative efficiency, postoperative cognition, and functional recovery.

Hypotheses: Patients in the VR group will have shorter post-anaesthesia care unit (PACU) length of stay as compared to sham VR + usual care controls. The effect of VR on postoperative delirium, postoperative cognitive decline, postoperative opioid use and functional recovery will be exploratory endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 60 or older undergoing primary total knee replacement surgery at BIDMC and receiving spinal/regional anesthesia
* English or Spanish speaking patients

Exclusion Criteria:

* Complex or revision surgeries
* Patients scheduled for "same day" TKA
* Open wounds or active infection of the face or eye area
* History of seizures or other symptom linked to an epileptic condition
* Patients who plan to wear hearing aids during the procedure
* Patients with a pacemaker or other implanted medical device
* Droplet or airborne precautions (as determined by local infection control policy)
* Non-English speaking or Non-Spanish speaking
* Moderate to severe dementia

Drop-Out Criteria:

* MoCA <10 (this test will be administered on Day of Enrollment)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Propofol Dose | Duration of the procedure, on average 1 to 3 hours
  Total propofol dose (mg/kg/min) administered intraoperatively

SECONDARY OUTCOMES:
Intraoperative and Postoperative Opioids | Duration of the procedure, on average 1 to 3 hours, and up until 72-hours postoperatively
  Total intraoperative and postoperative opioid equivalent doses administered
Intraoperative Anesthesia Maneuvers | Duration of the procedure, on average 1 to 3 hours
  Assessment of intraoperative vital signs and anesthesia maneuvers potentially related to over-sedation (i.e. airway interventions, use of airway assist devices, conversion to general anesthesia)
Length of PACU stay | Duration of the patient's stay in the post anesthesia care unit, on average 1 to 5 hours
  The length of the patients stay in the Post Anesthesia Care Unit.
Postoperative Pain | Measured on postoperative day zero and one, starting with PACU scores
  Clinically documented pain scores will be recorded on a scale from 0 (best outcome) to 10 (worst outcome). Using this numeric rating scale, patients will be asked to describe both the maximum and average level of pain
Satisfaction with Anesthesia | Within an hour of admission to the postoperative anesthesia care unit
  Patients will rate their overall satisfaction with their perioperative anesthesia care using the Iowa Satisfaction with Anesthesia Scale. They will also be asked to rate their satisfaction with their communication with their anesthesia providers.
Satisfaction with Recovery | Postoperative day one
  Patients will rate their overall satisfaction with their recovery from surgery using the QOR15. Additionally, patients will be asked how frequently they find themselves reacting to pain.
Postoperative Delirium | Measured daily on each postoperative day, starting on postoperative day 1 until postoperative day 7.
  A member of the research staff will meet with the patient and complete the 3-Minute Diagnostic Confusion Assessment Method (3D-CAM) to assess the incidence of postoperative delirium.
Delayed Cognitive Recovery and Postoperative Neurocognitive Disorder | Assessment will take place on day of enrollment and then at one week (+/- 48 hours) and one month postoperatively (+/- 7 days).
  Cognitive function will be assessed using the telephonic version of the Montreal Cognitive Assessment (MoCA).
Assessment of Knee Pain and Function | Assessments will take place within 7 days of the initial clinic visit and within 7 days of the initial postoperative clinic visit, typically one month after surgery.
  As part of standard pre and post TKA assessment, patients will be administered the Knee Injury and Osteoarthritis Outcome Score for Joint Replacement Patient-Reported Outcome Measures (KOOS-JR PROM) to assess the degree of limitation in activity and pain from their knee ailment.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P O'Gara, MD,MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Espinosa-Leon JP, Mathura R, Chen G, Joseph M, Sadhwani T, Beydoun N, Hernandez ER, Riley T, Kunze LJ, Goodspeed V, O'Gara BP. Intraoperative virtual reality for older patients undergoing total knee arthroplasty: study protocol for a randomized clinical trial. Trials. 2024 Dec 18;25(1):830. doi: 10.1186/s13063-024-08551-6. PMID 39695824